CLINICAL TRIAL: NCT02914496
Title: "Diabetes in Balance" - a Randomized Controlled Trial to Evaluate the Effects on Glucose Control, Self-care and Psychosocial Factors?
Brief Title: ACT Stress Management in Type 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Toft, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EPN Stockhom 2016/14-31/1
Record Dates: First submitted 2016-09-15; First posted 2016-09-26 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes in Balance (Experimental): The intervention consists of the manual-based CBT-group intervention "Diabetes in Balance". It is given in a group format with six to ten participants and consists of 7 sessions. The sessions are given bi-weekly for two hours. Each session has a specific theme such as "Stress and acceptance" "The life-compass; what is important in my life". The participants also conduct assignments related to the themes between the sessions. A licensed psychologist specialised in CBT and a diabetes specialist nurse, both trained in "ACT-stress management" will be leading the intervention group.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Control (No Intervention): The control group receives regular care including regular visits at the out-patient clinic, 3-4 times per year.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT is a specific form of Cognitive behavior therapy (CBT) which will be given as a course consisting of seven sessions where each session is two hours long.
  Other Names: Diabetes in Balance
  Arms: Diabetes in Balance

SUMMARY:
For many people living with type 1 diabetes it is a challenge to achieve good glucose control. Barely 20% reaches the goal level and many people experience self-care as complex, demanding and stressful. The purpose of this study is to evaluate the effect of a stress-management program on glucose control, self-care and psychosocial factors. The program is based on Acceptance and Commitment Therapy (ACT), a specific form of Cognitive behavior therapy (CBT). A total of 70 adult patients with type 1 diabetes from Ersta hospital will be recruited. Half of them will receive the intervention and the other half will continue with their regular diabetes care. A licensed psychologist specialised in CBT and a diabetes specialist nurse will be leading the intervention that is given in a group format. The program consists of seven 2-hour sessions given over 14 weeks. Glucose control, self care and stress will be measured at inclusion, after session four and seven, at six , 12 and 24 months and finally after 5 years

DETAILED DESCRIPTION:
ACT-stress management in type 1 diabetes - a randomized controlled trial to evaluate the effect on glucose control, self-control and psychosocial factors.

Purpose of proposed investigation:

The project hypothesis are that the CBT-intervention will a) improve glucose control, self-care, quality of life and acceptance of diabetes related thoughts and emotions and b) decrease depression, anxiety, general and diabetes related distress and fear of hypoglycemia.

Background information for the project:

The overall goal of diabetes management is to achieve good glycemic control while still maintaining good quality of life and experiencing as few hypoglycemic episodes as possible (the Swedish Social Board of Welfare, 2010). Currently only 19% of people with diabetes reach the goal of 52 mmol/mol for glycemic control (National Diabetes Registry, 2014). Research has proposed difficulties with behavior change (Knight et al., 2006), diabetes related distress (van Bastelar et al., 2010, Fisher et al., 2010) and fear of hypoglycemia (Wild et al., 2007) as important obstacles in achieving the goal. Patient education plays an important role in diabetes care but may not be sufficient in order to reach the recommended treatment goals. The association between knowledge and behavior change is weak and research has suggested that interventions should be more behavior oriented (Knight et al., 2006, Funnell et al., 2008). It is well known that people with chronic disease have an increased risk of developing psychological problems, for instance there are studies showing up to four times higher prevalence of depression in people with type 1 diabetes (Roy & Lloyd, 2012). It is also known that psychological problems are associated with poorer glycemic control, health and quality of life in this group (Chiechanowski et al., 2000; Jacobson, 2004).

Therefore, it is urgent to quickly discover and treat psychological problems. There is scientific support for Cognitive Behavior Therapy (CBT) to be effective in treating different types of anxiety (Stewart & Chambless, 2009) and depression (Cuijpers et al., 2011).

In light of this, different CBT-based interventions have been suggested as promising alternatives in treating diabetes. Several programs based on CBT have also been scientificly evaluated. Some of these studies have focused on changing concrete every day behaviors in order to promote self-care, glycemic control and quality of life (Snoek et al., 2008, Amsberg et al., 2009a,b) and some to treat co-morbid depression (Lustman et al., 1998). Our previous intervention study in this field (Amsberg et al., 2009 a, b) was the first one to show significant positive effects on glycemic control. In recent years a new form of CBT, Acceptance and Commitment Thearpy, (ACT), (Hayes, Strosahl, & Wilson, 1999) has received scientific attention. Of particular interest is that relatively short ACT-interventions in several studies have shown good results in a wide variety of psychosocial problems, smoking cessation, work related stress, anxiety, depression, chronic pain, epilepsi (Hayes et al., 2006).

" ACT-stressmanagement" is an intervention originally developed for preventing work-related stress and illness (Bond & Bunce, 2003) that later has been modified for different groups of peopel such as high-school students (Livheim, 2004), social workers (Brinkborg et al., 2011), medical students (Andersson & Waller, 2011). The intervention is designed so that different types of professionals, not only psychologists, can serve as group-leaders after a short period of training.

Plan of investigation:

The intervention "ACT-stress-management" will in this study be given as a course consisting of seven sessions where each session is two hours long. The course has been modified for people with diabetes so that the excercises and information will be related to diabetes and diabetes related problems. The sessions will be held every other week. The groups will consist of between six to a maximum of ten participants.

Subjects Inclusion criteria will be all adult (18-70 years) type 1 diabetes patients with HbA1c > 60 mmol/mol registered at Ersta hospital, diabetes- and endochrinology department/unit. The patient must be able to read, write and speak Swedish. Those with severe psychiatric conditions such as psychosis, recurrent severe depression or post-traumatic stress disorder, those with an ongoing cortison treatment, with co-morbid severe illness that affects glycemic control or are pregnant will be excluded.

Power-calculation:

A total of 56 patients (28 in the intervention group and 28 in the control group) are needed to achieve 80% power to detect the clinically relevant decrease of 6 mmol (The Association of Physical Activity, 2015) in HbA1c with 5% significance level and an SD of 9 mmol. In order to take in account of a drop-out rate of 24 % (Amsberg et al., 2008) during the study a total of 70 patients are needed to be included. The power-calculation was done with a web-based power-caculator.

Procedure:

The study consists of five main steps: 1. Recruitment of participants 2. The intervention 3. Psychometric evaluation of the Swedish version of AADQ 4. Data-processing 5. Presentation of the results

1. Recruitment of participants We will recruit a total of 70 patients during 2-3 years, of which half will receive the "ACT-stress-management" program and half will continue with treatment as usual. Patients fulfilling the inclusion criteria will meet the person collecting the data at the diabetes-center in order to receive information of the study and will at the same time be asked to participate in the study. At this time the participants will be informed orally and in writing about the study, recieve information about their possibility to leave the study at any time without any consequences, how data will be handled and finally about receiving a compensation in the form of a gift voucher of 100 SEK after each time they complete a set of questionnaires.
2. The intervention The intervention consists of: "The ACT-stressmanagement" intervention and administrating pre-intervention measurements, processmeasurments, post-intervention measurements and follow-up measurements. The control-group will only consist of the pre-, process-, post and follow-up measurements.

The intervention-group:

1. Informed consent for the study
2. After agreeing to being included, participants complete the set of questionnaires for base-line measures
3. "the ACT-stressmanagement" is given, including two process-measurements of AADQ
4. Post-intervention measurments
5. 1-year post inclusion follow-up measurements
6. 2-year post inclusion follow-up measurements
7. 5- year post inclusion follow-up measurements

The control-group:

1. Informed consent for the study
2. After agreeing to being included, participants complete the set of questionnaires for base-line measures
3. Treatment as usual, including two process-measurements of AADQ
4. Post-intervention measurments
5. 1-year post inclusion follow-up measurements

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Duration of disease >2 years -
* Hb1c>60 mmol/mol

Exclusion Criteria:

* Insufficient knowledge to understand and express themselves in Swedish
* Untreated or severe ongoing psychiatric disease
* Cortisone treatment
* Untreated thyroid disease
* Insulin pump therapy started since <3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 months post inclusion
  Measure of long term glucose control

SECONDARY OUTCOMES:
Manchester Short Assessment of Quality of life | 1-5 years post inclusion
  A form with 16 questions that examines the quality of life and satisfaction with life in general , employment, economy, friendships , leisure , housing , personal safety, and Health.
Depression Anxiety stress scales | 1-5 years post inclusion
  21 questions measuring depression, anxiety and stress during the last week.
The Hypoglycemia Fear Survey emotions, depression, anxiety, fear of hypoglycemia, general and diabetes related distress. | 1-5 years post inclusion
  A 23-items self-assessment questionnaire that appreciates concerns and behaviors in relation to hypoglycaemia.
The Problem Areas in Diabetes (Swe-PAID-20) Scale | 1-5 years post inclusion
  A questionnaire that measures the perception of burden in relation to diabetes and its treatment.
Acceptance and action diabetes questionnaire | 1-5 years post inclusion
  A questionnaire ( 11 questions ) that measures the emotional and cognitive avoidance related to diabetes.
The Summary of Self-Care Activities | 1-5 years post inclusion
  An instrument that reflects self-care activities such as SMBG, healthy eating and the implementation of optimal insulin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Anderbro, AssProf, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta sjukhus, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will primarily be presented at the group level. Individual data will where appropriate be anonymised

REFERENCES:
- [Derived] Wijk I, Amsberg S, Johansson UB, Livheim F, Toft E, Anderbro T. Impact of an Acceptance and Commitment Therapy programme on HbA1c, self-management and psychosocial factors in adults with type 1 diabetes and elevated HbA1c levels: a randomised controlled trial. BMJ Open. 2023 Dec 14;13(12):e072061. doi: 10.1136/bmjopen-2023-072061. PMID 38101850
- [Derived] Amsberg S, Wijk I, Livheim F, Toft E, Johansson UB, Anderbro T. Acceptance and commitment therapy (ACT) for adult type 1 diabetes management: study protocol for a randomised controlled trial. BMJ Open. 2018 Nov 28;8(11):e022234. doi: 10.1136/bmjopen-2018-022234. PMID 30498037